CLINICAL TRIAL: NCT06693947
Title: A Pilot Study in the Swiss Alps: Impact of Alpine Dairy Products on Blood Lipid Levels
Brief Title: Impact of Alpine Dairy Products on Blood Lipid Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Fribourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-01411
Record Dates: First submitted 2024-09-26; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Elevated Cholesterol
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alpine dairy products (Experimental): Intake of 3 portions of alpine dairy products made from milk of cows grazing in subalpine to alpine regions in the Swiss alps in Val Müstair (GR) (one portion equals 2 dl milk, 150-200 g yoghurt, quark, cottage cheese, other dairy products, 30g hard cheese, 60g soft cheese) during the 6-week intervention period. Every dairy product intake will be reported into the participants' food log. Participants will be instructed not to change their diet (with the exception of dairy products), lifestyle and physical activity during the study.
  Interventions: Other: Alpine dairy products
- Non-alpine dairy products (No Intervention): Intake of 3 portions of standard dairy products made from milk of cows grazing in lower altitudes, found in local food stores, thus avoiding alpine dairy products during the 6-week intervention period. There are no other restrictions, all dairy products are considered equivalent. Every dairy product intake will be reported into the participants' food log. The participants will be instructed not to change their diet (with the exception of dairy products), lifestyle and physical activity during the study.

INTERVENTIONS:
Other: Alpine dairy products — The intervention group will be instructed to eat three portions of alpine dairy products daily. The proposed three portions represent an estimated mean consummation in the study population, taking into consideration the national statistics.
  Arms: Alpine dairy products

SUMMARY:
Elevated blood lipid levels are one of the main risk factors for cardiovascular disease. To manage elevated blood lipid levels in otherwise healthy people at low risk of cardiovascular disease, lifestyle changes are recommended as the first treatment strategy. One of these changes concerns diet. Clinical observations by general practitioners in alpine regions of Switzerland have shown that consumption of dairy products produced from cows living and grazing at high altitudes can have a beneficial effect on blood lipid parameters. However, little clinical data is available on the effect of alpine dairy products on health-related markers. This pilot study aims to assess if replacing standard (non-alpine) dairy products by alpine dairy products in the daily diet among patients with elevated LDL-cholesterol levels could reduce the blood LDL-cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Elevated lipid levels, namely: fasting LDL-cholesterol >3mmol/L and </=5mmol/L
* Agreeing to eat 3 portions of dairy products daily (according to instructions)

Exclusion Criteria:

* Eating less than two and more than six portions of dairy products daily
* Body weight change +/-5% of body weight in the last three months
* Secondary prevention treatment for cardiovascular disease
* Moderate, high or very high cardiovascular risk according to AGLA score
* Currently taking PSCK9-inhibitors, ezetimibe, statins, glucocorticoids
* Poorly controlled, severe chronic renal insufficiency, hypothyroidism, cholestasis, nephrotic syndrome, eating disorders, alcohol abuse, Cushing syndrome
* Myocardial infarction, percutaneous coronary intervention or coronary artery bypass grafting in the previous 6 months
* Known lactose intolerance or dairy allergies
* Change of diet less than 2 months before intervention
* Pregnant or breastfeeding
* Incapacity of judgement
* Inability to speak and read German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Change in fasting blood LDL-cholesterol level | Baseline, Day 15, Day 30 and Day 45
  Measure of LDL-cholesterol in mmol/L

SECONDARY OUTCOMES:
Change in total cholesterol, triglycerides, HDL-cholesterol and lipoprotein A | Baseline, Day 15, Day 30 and Day 45
  Measures in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Rodondi, Prof, Study Director — University of Fribourg
Locations (1):
- Center da Sandà Val Müstair, Santa Maria, Switzerland

IPD SHARING:
Plan to Share IPD: No